CLINICAL TRIAL: NCT00792012
Title: A Phase I Dose Per Fraction Escalation Study of Hypofractionated Intensity-Modulated Radiation Therapy (Hypo-IMRT) Combining With Temozolomide (TMZ) Chemotherapy for Patients With Newly Diagnosed Glioblastoma Multiforme (GBM)
Brief Title: A Dose Per Fraction Escalation Trial of Hypofractionated IMRT With Temozolomide for Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0562.cc
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glioblastoma Multiforme Patients (Experimental): Hypofractionated Intensity-Modulated Radiation Therapy (Hypo-IMRT) Combining with Temozolomide (TMZ) Chemotherapy
  Interventions: Radiation: Hypofractionated Intensity-Modulated Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Radiation: Hypofractionated Intensity-Modulated Radiation Therapy — All patients will receive one fraction of radiation therapy a day, 5 days a week, Monday through Friday. Radiation fraction size and number of fractions depend on dose fraction level the patient is assigned to.
Drug: Temozolomide — Temozolomide will be administered orally, once a day starting on the first day of radiation, for 28 consecutive days during radiation, and after radiation for those patients completing radiation in less than 28 days.
  Other Names: Temodar

SUMMARY:
The purpose of the study is to find out the highest dose per fraction of hypofractionated Intensity-Modulated Radiation Therapy (Hypo-IMRT) that can be safely given with temozolomide chemotherapy.

DETAILED DESCRIPTION:
Hypo-IMRT is given in fewer treatments than conventional radiation therapy. This will be a dose per fraction escalation study. A dose per fraction escalation study means that successive groups of patients will receive higher doses per fraction of radiation while keeping the total dose of radiation the same (60 Gy, Gy is a radiation unit). The radiation dose per fraction will be increased and the numbers of radiation treatments will be decreased until a fraction dose is reached at which there are unacceptable side effects compared with possible benefit. Which group subjects are assigned to will depend on what stage the study has reached at the time the subject decide to participate.

This research is being done because with current standard radiation therapy (A total dose of 60 Gy given 2 Gy a day over 6 weeks) the outcome is very poor. New and more effective radiation therapy methods are desperately needed for patients with GBM.

In this study, radiation therapy is given together with chemotherapy of Temozolomide.

This study is also designed to monitor the level of some of the known cytokines (specific proteins in the blood) before and after radiation, and in meantime to screen unknown proteins in patients' blood before and after radiation therapy. Hopefully, this will provide some clues for future study of monitoring radiation damage, and possibly new therapeutic approach for patients with GBM.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed WHO grade IV astrocytoma (GBM), tumor can be supra- or infra-tentorial in location but not located in the brain stem.
* Solitary or multifocal tumor.
* Tumor can be biopsied or resected, either totally or sub-totally.
* A pre-radiation therapy brain MRI is mandatory.
* Surgical cavity or surgical cavity + T1 enhancing residual tumor ≤ 6 cm in the largest diameter on the pre-radiation therapy MRI. In the case of multifocal tumor, the combined largest diameter of T1 enhancing tumor + surgical cavity ≤ 6 cm.
* Placement of bis-chloronitrosourea (BCNU) wafers at the time of surgery is allowed.
* Age > 18 years at time of registration.
* Estimated survival of at least 3 months.
* Zubrod Performance Scale of 0-2 (Karnofsky performance scale ≥ 60).
* Hgb > 9 gm; absolute neutrophil count (ANC) > 1500/ul; platelets > 100,000; Creatinine < 1.5 times the upper limit of laboratory normal value; Bilirubin < 2 times the upper limit of laboratory normal value; serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) < 3 times the upper limit of laboratory normal value.
* Patients must sign study-specific informed consent form prior to registration.
* Men and women and members of all ethnic groups are eligible for this trial.
* Radiation therapy and chemotherapy must start within 8 weeks of tumor resection or biopsy

Exclusion Criteria:

* Patients with contraindications for MRI scanning.
* Prior temozolomide chemotherapy.
* Prior brain irradiation.
* Evidence of severe or uncontrolled psychiatric or systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) that would interfere with study protocol as judged by the investigator.
* Acquired Immune Deficiency (HIV (+)/AIDS)
* Patients being treated on any other clinical protocols within 30 days prior to study entry or during participation in the study.
* Pregnant women or breast feeding women. Women of childbearing potential must practice medically approved contraceptive precautions. Men should be counseled and agreeable to follow acceptable birth control methods.
* Active connective tissue disorders, such as active lupus or scleroderma.
* Concurrent active malignancy at other sites.
* Frequent vomiting of medical condition which could interfere with oral medication intake (e.g. partial bowel obstruction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To identify the maximum dose per fraction of IMRT a patient can tolerate while keeping the total radiation dose at 60 Gy, provided concurrently with daily oral temozolomide chemotherapy | Up to 60 days
  To determine the frequency of patients developing >= grade 3 acute and delayed toxicities attributable to radiotherapy. Acute radiotherapy toxicities are defined as those toxicities which occur during and within 30 days from the completion of radiotherapy and delayed toxicity are those developed at least 30 days after the last dose of radiation.

SECONDARY OUTCOMES:
Progression-free survival | Until disease progression
  To monitor the level of some of the known and unknown cytokines or proteins before and after Hypo-IMRT and correlate it with the incidence of acute and late neurotoxicity. Quality of life assessment before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Ney, M.D, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy K, Damek D, Gaspar LE, Ney D, Waziri A, Lillehei K, Stuhr K, Kavanagh BD, Chen C. Phase II trial of hypofractionated IMRT with temozolomide for patients with newly diagnosed glioblastoma multiforme. Int J Radiat Oncol Biol Phys. 2012 Nov 1;84(3):655-60. doi: 10.1016/j.ijrobp.2012.01.035. Epub 2012 Apr 5. PMID 22483738